CLINICAL TRIAL: NCT04202939
Title: nutritionDay in Nursing Homes: An International Audit and Registry on Nutrition and Outcome
Brief Title: nutritionDay in Nursing Homes Worldwide: An International Audit and Registry on Nutrition and Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: European Society for Clinical Nutrition and Metabolism (Other); Austrian Society for Clinical Nutrition (Other)
Responsible Party: Principal Investigator, Michael J. Hiesmayr, Professor of Anesthesia and Intensive Care, Medical University of Vienna
Other Study IDs: 407/2005 (nursing homes)
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status; Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- nursing homes residents: all residents present in a nursing home unit on nutritionDay
  Interventions: Other: nutrition

INTERVENTIONS:
Other: nutrition — type and amount of food eaten or type of oral nutritional supplements as well as enteral or parenteral nutrition
  Other Names: nursing home food; oral protein energy supplements; enteral nutrition; parenteral nutrition

SUMMARY:
Due to longer life expectancy, age-related changes and problems become more significant. The aging process is associated with loss of function and reduced performance. Age-related physiological changes in the regulation of nutrition intake and in the gastro-intestinal tract lead to deterioration of the nutritional status. Deterioration of the health status and of nutritional intake is further associated with chronic malnutrition, impaired quality of life, increased morbidity, mortality and long-term care. In order to ensure optimal nutritional care of nursing home residents and therefore have a lasting positive affect on their quality of life, morbidity and mortality, it is necessary:

* to collect data on the quality of nutritional care in nursing homes by means of a simple method that requires no specialization in data acquisition,
* to acquire knowledge on the prevalence of risk factors of malnutrition in nursing home residents in general and on individual nursing units, also in conjunction with the outcome after six months, and to forward the same to the individual nursing units,
* to allow comparison with other facilities (with similar profile) with the help of a benchmarking system,
* to assess the effectiveness of introduced changes in terms of quality management and quality improvement.

DETAILED DESCRIPTION:
The study is a population-based, observational cross-section examination carried out on one day, and an outcome evaluation six months later. The examination should be repeated annually. Data is collected with the help of questionnaires. Anonymised data entry into the audit database is done with individual and anonymous center and unit-codes.

There are 2 questionnaires to complete on nutritionDay. The unit staff completes 1 questionnaire about structure of the unit and 1 questionnaire about resident characteristics.

1. unit sheet: asks for nutrition related organisational and structural information on the unit.
2. resident description: asks for general characteristics, diseases, care level, mobility and restrictions on food intake.

Outcome Evaluation: re-assesses the resident's outcome 6 months after nutritionDay (residence after 6 months, actual weight, and hospitalization). This questionnaire has to be completed 6 months after nutritionDay by the unit staff.

Participation rules:

1. A user needs to register to nutritionDay as a member to the nutritionDay network. Each may choose a personal user name. Each user needs to provide a valid email address. After responding to a validation email the user is registered with the chosen user name. User details are stored on a system that is not connected to the nutritionDay registry at any time. One user may serve as contact for several units and centers.
2. A user may order codes for participation for one or several centers and units. Access to the registry is only possible with a center code and unit code. These codes are selected from a list of random numbers.

Audit/registry recruitment plan:

Participation to the registry is voluntary. There is actually no participation fee. All necessary information can be obtained from a dedicated website (www.nutritionday.org). Participation can be promoted via international and national scientific societies, universities, health care organisations or governmental agencies as well as via advertisement at international and national congresses. T

Risk and benefit assessment:

The study implies no risk whatsoever for the residents. On some levels participation can even be expected to be beneficial:

* Direct benefit for residents through increased attention to nutritional problems.
* Raising awareness of decision-makers brought about by the decision-making process taking place prior to participating in the study and receiving the quality report of the nursing unit or facility.
* Increase awareness of the staff of nursing homes by participating in the study and the quality report. Pilot results suggest that in terms of the Hawthorne effect, just participation alone has a positive influence on nutrition management on nursing units.
* Since the project is planned for at least two years, it is possible to repeat the study after one year, to be able to monitor changes which were introduced as a result of the first report.
* Due to prior announcement on the nursing units, residents and their trustees are made aware of the issue of malnutrition and proper diet management. The nutritionDay in hospitals has shown that in many cases for the first time discussions between staff, patients and relatives on this subject were set in motion.

Documentation of the results of the study, data management and data security

All the necessary data for documentation of the study are entered on the questionnaires. On the study forms the nursing unit is identified by a numerical code, which is allocated after application from the audit facility. The questionnaires only include information on year of birth of the residents and their initials. If requested by the nursing units, to facilitate the evaluation of outcomes. the evaluation can be completed without the initials.

The data are entered online into the database from the facility. The coordination center does not have access at any time to documents that would influence the anonymity of the residents.

The data in the coordination center is checked for credibility prior to further evaluation. In the case of unclear or incomplete data, feedback to the responsible person on the nursing unit takes place and a possible correction of data is made. All data are analyzed anonymously, and the results are made available to each nursing unit so that the identity of the nursing unit, as well as the anonymity of the individual residents is assured.

Communication of Results Following data input of the resident's outcome, each nursing unit (the nutritionDay Project Leader person on the ward nursing unit responsible for organizing the nutritionDay and should be who is clearly identifiable by an e-mail address) receives the results compared to the whole project in the form of a quality report on nutritional intake and influencing factors.

The results of the study are published by the head of the study in a scientific journal and presented at scientific conferences.

Statistical Methods An analysis on survival with the target variable "death in nursing homes within six months" will be carried out. Existing risk factors are to be taken into account as covariant causes. Information on the time of admission to the nursing home and the time of death of the residents will be available.

In addition, the trend of weight development of the surviving residents between the nutritionDay and a half year thereafter will be recorded. The connection between nutritional status and weight on the nutritionDay and the course of weight thereafter of the surviving residents will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* nursing home resident
* minimum age: 50
* present on nursing home unit on nutritionDay

Exclusion Criteria:

* 49 years and under
* resident refused to participate in nutritionDay

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study evaluates nursing homes units and their residents who must be 50 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2007-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dependence of nutritional intake on nutritional status and risk factors | 180 days
  dependence of the outcome of nursing home residents' on their nutrient intake, their current nutritional status and risk factors (state of health, level of care

SECONDARY OUTCOMES:
Nutrition-related structural parameters | 180 days
  structural parameters (number and type of unit staff, implementation of regular nutrition screening

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hiesmayr, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upon submission of a research proposal data anonymised data are shared with researcher. Each proposal is submitted to the supervisory board for approval.

REFERENCES:
- [Background] Streicher M, Wirth R, Schindler K, Sieber CC, Hiesmayr M, Volkert D. Dysphagia in Nursing Homes-Results From the NutritionDay Project. J Am Med Dir Assoc. 2018 Feb;19(2):141-147.e2. doi: 10.1016/j.jamda.2017.08.015. Epub 2017 Oct 10. PMID 29030310
- [Background] Streicher M, Themessl-Huber M, Schindler K, Sieber CC, Hiesmayr M, Volkert D. nutritionDay in Nursing Homes-The Association of Nutritional Intake and Nutritional Interventions With 6-Month Mortality in Malnourished Residents. J Am Med Dir Assoc. 2017 Feb 1;18(2):162-168. doi: 10.1016/j.jamda.2016.08.021. Epub 2016 Oct 11. PMID 27742584
- [Background] Streicher M, Themessl-Huber M, Schindler K, Sieber CC, Hiesmayr M, Volkert D. Who receives oral nutritional supplements in nursing homes? Results from the nutritionDay project. Clin Nutr. 2017 Oct;36(5):1360-1371. doi: 10.1016/j.clnu.2016.09.005. Epub 2016 Sep 17. PMID 27692932
- [Background] Wirth R, Streicher M, Smoliner C, Kolb C, Hiesmayr M, Thiem U, Sieber CC, Volkert D. The impact of weight loss and low BMI on mortality of nursing home residents - Results from the nutritionDay in nursing homes. Clin Nutr. 2016 Aug;35(4):900-6. doi: 10.1016/j.clnu.2015.06.003. Epub 2015 Jun 19. PMID 26143743
- [Background] Valentini L, Schindler K, Schlaffer R, Bucher H, Mouhieddine M, Steininger K, Tripamer J, Handschuh M, Schuh C, Volkert D, Lochs H, Sieber CC, Hiesmayr M. The first nutritionDay in nursing homes: participation may improve malnutrition awareness. Clin Nutr. 2009 Apr;28(2):109-16. doi: 10.1016/j.clnu.2009.01.021. Epub 2009 Mar 5. PMID 19264381
- See also: nutritionDay project website — https://www.nutritionday.org/